CLINICAL TRIAL: NCT05801796
Title: Analyzing Factors of Patient Involvement in Ovarian Cancer Clinical Trials
Brief Title: Appraising Medical Trial Experiences of Ovarian Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 89480700
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical trials has been highly skewed towards specific demographic groups. However, research identifying which trial attributes impact participation, in either positive or negative ways, is limited. This study invites participants to record a wide range of data on their clinical trial experience, with the goal being to identify factors which persistently limit patients' ability to participate in, or complete, a trial in which they were initially interested. Data will be analyzed through a range of demographic lenses, in hopes of discovering patterns which might improve the experience of future ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Patient has been diagnosed with ovarian cancer
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form
* Pregnant, breastfeeding or expecting to conceive within the projected duration of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Ovarian cancer patients who are actively considering enrolling in a medical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient decides to enroll in clinical trial | 3 Months
Patient remains in clinical trial to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cho KR, Shih IeM. Ovarian cancer. Annu Rev Pathol. 2009;4:287-313. doi: 10.1146/annurev.pathol.4.110807.092246. PMID 18842102
- [Background] Eisenhauer EA. Real-world evidence in the treatment of ovarian cancer. Ann Oncol. 2017 Nov 1;28(suppl_8):viii61-viii65. doi: 10.1093/annonc/mdx443. PMID 29232466
- [Background] Previs RA, Secord AA. Ovarian Cancer: Clinical Trial Breakthroughs and Impact on Management. Obstet Gynecol Clin North Am. 2019 Mar;46(1):67-88. doi: 10.1016/j.ogc.2018.09.005. PMID 30683267

DOCUMENTS (1):
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT05801796/ICF_000.pdf